CLINICAL TRIAL: NCT01363167
Title: Identifying Vit D Deficiency in VLBW Infants Part 2
Brief Title: Identifying Vitamin D Deficiency in Very Low Birth Weight Infant (VLBW) Infants Part 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Principal Investigator, Sarah N Taylor, Assistant Professor of Pediatrics, Medical University of SC, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HR# 17217; K23RR021891 (NIH)
Record Dates: First submitted 2011-04-18; First posted 2011-06-01 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2014-11

CONDITIONS: Infant, Very Low Birth Weight; Calcium Deficiency; Vitamin D Deficiency
Keywords: vitamin D; preterm infants; calcium; bone; parathyroid hormone
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 400 IU Cholecalciferol - Vitamin D (Active Comparator)
  Interventions: Dietary Supplement: 400 IU Cholecalciferol- Vitamin D Daily
- Placebo (Placebo Comparator): Placebo contains Fractionated Coconut Oil
  Interventions: Dietary Supplement: 400 IU Cholecalciferol- Vitamin D Daily

INTERVENTIONS:
Dietary Supplement: 400 IU Cholecalciferol- Vitamin D Daily — Infants who are defined as vitamin D deficient at birth will be randomized to receive either 400 IU vitamin D/day or placebo daily until term age is reached.

SUMMARY:
This study is to determine the amount of vitamin D required for a very low birth weight infant to reach vitamin D sufficiency and achieve optimal calcium health and bone growth.

ELIGIBILITY:
Inclusion Criteria:

* Any infant born at the Medical University of South Carolina <34 weeks gestation
* Less that 1500g at birth
* AGA
* Must be African American or Caucasian
* Each infant born of twin and triplet pregnancies will be eligible

Exclusion Criteria:

* Infants with major congenital anomalies or with hemolytic disease requiring exchange transfusion
* Infants born small for-gestational-age (SGA) or large for-gestational-age (LGA)
* Maternal uncontrolled thyroid disease
* Maternal Parathyroid disease
* Infants of races other than African American or Caucasian

Ages: 1 Day to 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68 (Actual)
Dates: Start 2011-10; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Intestinal Calcium Absorption | When receiving at least 50% of nutrition enterally expected to occur at 2-6 weeks post-birth
Parathyroid hormone concentration | At term age (expected 2-4 months)
Serum 25 hydroxyvitamin D status | At term age (expected 2-4 months)
Bone Health | At term age (expected 2-4 months)
  Bone ultrasound measurement, serum alkaline phosphatase, and bone-specific alkaline phosphatase at birth and monthly until term age. Bone mineralization by DEXA scan at hospital discharge and term age.
Serum inflammatory cytokine concentrations | At birth (day 1)

SECONDARY OUTCOMES:
Phosphorus Homeostasis | At term age (expected 2-4 months)
  Measurement of serum and urine phosphorus concentrations
Growth parameters | At term age (expected 2-4 months)
Vitamin D Dose Safety as Measured by Urinary Calcium Excretion | At term age (expected 2-4 months)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah N. Taylor, M.D., Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States